CLINICAL TRIAL: NCT00327392
Title: A Phase 3 Open-Label, Single Arm Study to Assess the Safety of AQUAVAN® (Fospropofol Disodium) Injection for Minimal-to-Moderate Sedation in Patients Undergoing Minor Surgical Procedures
Brief Title: A Safety Study of AQUAVAN® (Fospropofol Disodium) Injection for Sedation During Minor Surgical Procedures.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3000-0523
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Procedural Sedation
Keywords: Arthroscopy; AV Shunt; Bunion; Dilatation and Curettage; Esophagogastroduodenoscopy; Hysteroscopy; Lithotripsy; Rotator Cuff/ Shoulder; Transesophageal Echocardiography; Ureteroscopy; AQUAVAN; Sedation
MeSH Terms: conditions — Arteriovenous Fistula; Bunion; Dilatation, Pathologic | interventions — fospropofol; Injections

INTERVENTIONS:
Drug: AQUAVAN® (fospropofol disodium) Injection

SUMMARY:
Very often patients receive medications before a diagnostic, therapeutic, or surgical procedure to help them relax, keep them calm, and to relieve them from pain. This is called procedural sedation. With respect to minimal-to-moderate procedural sedation for minor surgical procedures, a patient is first given a pain-relief medication (analgesic) and then a medication to help him/her relax and keep calm (sedative). AQUAVAN is a chemically modified form of propofol, a commonly-used sedative drug. AQUAVAN acts like a slow release version of propofol, and is being studied to see if it can safely keep patients calm and relaxed during their medical procedure and then allow for rapid and clear-headed recovery.

DETAILED DESCRIPTION:
This is a Phase 3 open-label, single-arm study designed to evaluate the safety of AQUAVAN following pretreatment with an analgesic, fentanyl, in patients who are undergoing minor surgical procedures that require minimal-to-moderate sedation. All patients will be placed on supplemental oxygen via nasal cannula and an electrocardiogram monitor, pulse oximeter, and blood pressure monitor will be attached prior to administration of fentanyl. Assessments will be made to evaluate the safety of AQUAVAN in patients undergoing minor surgical procedures.

ELIGIBILITY:
- Number of sites/patients: Approximately 18 sites and 125 patients.

Inclusion Criteria:

1. Patient must be able to understand, either orally or in writing, and be able to consent and complete the required assessments and procedures.
2. Patient provides signed/dated Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) of 1996 authorization after receiving a full explanation of the extent and nature of the study.
3. Patient must be at least 18 years of age and undergoing one of the specified minor surgical procedures at the time of screening.
4. If female, patient must be surgically sterile, postmenopausal, or not pregnant or lactating and must have been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and predose.
5. Patient meets American Society of Anesthesiologists (ASA) Physical Classification System status of P1 to P4.

Exclusion Criteria:

1. Patient has a history of allergic reaction or hypersensitivity to any anesthetic agent or opioid.
2. Patient does not meet nils per os (NPO) status per ASA guidelines or institution's guideline.
3. Patient has a Mallampati Classification Score of 4; or a Mallampati Classification Score of 3 and a thyromental distance <4 cm, or for any other reason has a difficult airway, in the opinion of the Principal Investigator.
4. Patient has an abnormal, clinically significant 3-lead ECG finding at predosing period.
5. Patient has participated in an investigational drug study within 1 month prior to study start.
6. Patient is unwilling to adhere to pre- and postprocedural instructions.
7. Patient for whom the use of fentanyl citrate injection (fentanyl) is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-05; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Jones, MD, PharmD, Study Director — Eisai Inc.
Locations (15):
- United States (15):
  - Precision Trials, Phoenix, Arizona
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Louisville, Louisville, Kentucky
  - Medical Research Institute, Inc., Slidell, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - St. Louis Women's Healthcare Group, Chesterfield, Missouri
  - International Heart Institute of Montana, Missoula, Montana
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Carolina Urologic Research, Myrtle Beach, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - Physicians' Research Options, Sandy City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited at 12 study centers in the US during the period of 22-Jun-2006 to 01 Mar 2007.
Pre-assignment Details: All subjects received fentanyl at an initial dose of 50 μg as an analgesic pretreatment 5 minutes prior to the administration of the initial dose of fospropofol disodium (also referred to as LUSEDRA and formerly known as AQUAVAN). After fentanyl administration, the venous catheter was flushed with 2 mL of sterile saline solution.
Groups:
- Fospropofol Disodium: Fospropofol disodium 6.5 mg/kg (no less than 390 mg and no more than 585 mg, based on age, weight, and American Society of Anesthesiologists [ASA] Status): one initial intravenous (i.v.) bolus dose. Supplemental doses of fospropofol disodium 1.63 mg/kg (no less than 97.5 mg and no more than 146 mg) were administered as needed.
Period: Overall Study
Arm/Group | Fospropofol Disodium
Started | 123
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fospropofol Disodium
Number analyzed (Participants) | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 56
Race/Ethnicity, Customized [Number; unit: particpants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 109
  More than one race | 0
  Unknown or Not Reported | 0
  Hispanic/Latino | 3
  Other | 1
Weight (kg) [Number; unit: participants]
  <60 | 18
  >60 to <90 | 69
  >90 | 36
American Society of Anesthesiologists (ASA) status [Number; unit: participants]
  P1 ( A normal healthy patient ) | 33
  P2 ( A patient with mild systemic disease ) | 67
  P3 ( A patient with severe systemic disease ) | 22
  P4 (High risk, severely compromised by disease) | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Airway Assistance in Patients Undergoing Minor Surgical Procedures
Time Frame: 2 hours
Population: Number of patients requiring specified types of airway assistance
Measure: Number; unit: particpants
Arm/Group | Fospropofol Disodium
Number analyzed (Participants) | 7
particpants
  Verbal Stimulation | 1
  Loud Tone of Voice | 1
  Face Mask | 1
  Chin Lift | 1
  Oral Airway | 1
  Increased Oxgen Flow | 2

ADVERSE EVENTS:
Arm/Group | Fospropofol Disodium
Serious Adverse Events (participants affected / at risk) | 4/123
Other Adverse Events (participants affected / at risk) | 111/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fospropofol Disodium (N=123)
Cardiac arrest (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 2
Ammonia increased (Investigations) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fospropofol Disodium (N=123)
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 7
Procedural pain (Injury, poisoning and procedural complications) | 62
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Paresthesia (Nervous system disorders) | 66
Tremor (Nervous system disorders) | 2
Uterine spasm (Reproductive system and breast disorders) | 4
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 32
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No